CLINICAL TRIAL: NCT03551080
Title: Inflammation Och hjärnfunktion - Pilotstudie
Brief Title: Inflammation and Brain Function - Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: University of California, San Francisco (Other); The Swedish Society of Medicine (Other); Swedish Heart Lung Foundation (Other); The Swedish Research Council (Other Government); Swedish Council for Working Life and Social Research (Other); Stockholm University (Other)
Responsible Party: Principal Investigator, Mats Lekander, Professor, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2008/955-31
Record Dates: First submitted 2018-05-29; First posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Sickness Behavior
Keywords: Sickness behavior; Cytokines; Psychoneuroimmunology
MeSH Terms: conditions — Illness Behavior | interventions — Lipopolysaccharides; Endotoxins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endotoxin (Active Comparator): 0.8 ng lipopolysaccharide/kg body weight injection
  Interventions: Biological: Lipopolysaccharide
- Placebo (Placebo Comparator): Saline injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Lipopolysaccharide — Endotoxin at 0.8 ng/kg of body weight administered intravenously (Escherichia Coli, Lot nr G3E0609, United States Pharmacopeia Rockville, MD)
  Other Names: Endotoxin; LPS
  Arms: Endotoxin
Biological: Placebo — Saline administered intravenously
  Arms: Placebo

SUMMARY:
In this randomized double blind cross-over study 8 healthy persons were injected with 0.8 ng/kg body weight lipopolysaccharide (LPS) /endotoxin and placebo at two different occasions. The aim was to investigate how pain sensitivity and health perception change in response to an acute immune activation.

DETAILED DESCRIPTION:
Eight healthy participants were included in this randomized and balanced double blind cross-over study. They were injected two times, once with the active component and once with placebo. Participants were recruited by advertising and screened through questionnaires and a health examination by a physician. They were asked not to engage in strenuous physical activities, sleep regular hours and refrain from alcohol the day before the experiment. If the participants felt ill, e.g. coming down with a cold, they were instructed to call and were rescheduled for a later appointment. C-reactive protein (CRP) was assessed to exclude participants having an ongoing infection on the experimental day. Pregnancy was also an exclusion criteria and a pregnancy test was administered for all female participants on arrival. Several pain sensitivity measures were performed baseline and at peak inflammatory response 1-2 hours after injection. Subjects filled out questionnaires at baseline, 90 minutes and 4,5 hours after injection.

The study and the procedures used in the study are described in detail here: https://openarchive.ki.se/xmlui/bitstream/handle/10616/44650/Thesis_Bianka_Karshikoff.pdf?sequence=8&isAllowed=y

The following papers have been published using data from this study:

Olsson MJ, Lundstrom JN, Kimball BA, Gordon AR, Karshikoff B, Hosseini N, Sorjonen K, Olgart Hoglund C, Solares C, Soop A, Axelsson J & Lekander M. The Scent of Disease: Human Body Odor Contains an Early Chemosensory Cue of Sickness. Psychol Sci. 2014 Jan 22.

Sundelin T, Karshikoff B, Axelsson E, Hoglund CO, Lekander M, Axelsson J. Sick man walking: Perception of health status from body motion. Brain Behav Immun. 2015;48:53-6.

Karshikoff B, Lekander M, Soop A, Lindstedt F, Ingvar M Kosek E, Olgart Höglund C, & Axelsson J. Modality and sex differences in pain sensitivity during human endotoxemia. Brain, Behavior, and Immunity. 2015 May;46:35-43

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Diagnosed physiological or psychiatric disease
* Needle anxiety or blood phobia
* Regular medication (excluding contraceptive pill)
* Infection in the last two weeks
* Pregnancy or breastfeeding
* Smoking
* Excessive alcohol use
* Body mass index in the range of obesity (>30 kg/m2) or underweight (<18.5 kg/m2)
* Invisible veins in the antecubital area of the arms

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change in interoceptive vs exteroceptive focus | 7 hours
  Rating of concordance of heartbeat vs signal and change in tone of signal

SECONDARY OUTCOMES:
Change in self-rated health | 7 hours
  Two questions were used to assess self-rated health 1"how do you rate your general health status" rated on a 5 grade Likert scale very good to very poor and 2"how is your health right now" rated on a 7 grade Likert scale from excellent to very poor
Change in pain perception | 7 hours
  Both deep and cutaneous pain at threshold and suprathreshold noxious levels. Heat- and cold (cutaneous) pain sensitivity was assessed for threshold stimuli and intense noxious stimuli, as well as pressure (deep) pain thresholds and CPM (descending pain inhibition).
Change in facial apparence | 2 hours
  Photos were taken under standardised conditions before and after injection
Change in gait | 2 h
  The participants were filmed walking before and after injection

IPD SHARING:
Plan to Share IPD: Undecided